CLINICAL TRIAL: NCT05814289
Title: The Association of Telephone Head Tilt With Cervical, Thoracic, and Lumbar Spine Mobility and Disorders in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 83116987-712
Record Dates: First submitted 2023-03-16; First posted 2023-04-14 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-04

CONDITIONS: Forward Head Posture
Keywords: Head tilt; Lumbar spine; Spine; Cervical spine; Thoracic spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy young adults group (Other): To assess telephone head tilt and cervical, thoracic, and lumbar spine mobility and disturbances.
  Interventions: Other: To assess telephone head tilt and cervical, thoracic, and lumbar spine mobility and disturbances.

INTERVENTIONS:
Other: To assess telephone head tilt and cervical, thoracic, and lumbar spine mobility and disturbances. — To assess telephone head tilt and cervical, thoracic, and lumbar spine mobility and disturbances.

SUMMARY:
To determine the relationship between telephone head tilt and cervical, thoracic, and lumbar spine mobility and disturbances in young adults.

DETAILED DESCRIPTION:
Today, the fact that smartphones are easily portable and can be used for many purposes such as playing games, surfing the Internet, accessing information, shopping, and listening to music has made them widespread at an unexpected rate. This situation has brought the issue of device addiction to the agenda. Smartphone addiction can lead to many physical ailments such as visual impairment, numbness, and tingling in the hands, neck, back, hip, and knee pain. In the studies conducted, smartphone addiction was determined in university students and this situation was found to be associated with musculoskeletal pain. Considering the smartphone usage rates, durations, and smartphone usage postures of young adults, it can be predicted that spinal mobility may be adversely affected and may cause spine-related disorders. This study aims to determine the relationship between telephone head tilt and cervical, thoracic, and lumbar spine mobility, and disorders in young adults. In addition, it is aimed to examine the relationship between these parameters with quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Using smartphone,
* Not having any diagnosed chronic disease,
* No past or present mental illness,
* Individuals who can speak, read and write Turkish.

Exclusion Criteria:

* Having any neurological, psychiatric or cognitive disorder,
* Individuals who cannot speak, read or write Turkish.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Telephone head tilt | 1 day
  Telephone head tilts of individuals will be measured with a goniometer. Individuals will be asked to sit in the position where they use the phone in daily life. The cervical 7th Vertebra (C7) and tragus will be determined and the angle between them and the vertical line will be recorded in degrees. In order to reduce the error rate of the measurement, three evaluations will be made and averaged.
Cervical, Thoracic, and Lumbar Spine Mobility | 1 day
  Active range of motion for cervical, thoracic, and lumbar spine mobility will be measured with two bubble inclinometers (Baseline Bubble Inclinometer, White Plains, NY).
Core Outcome Measurement Index | 1 day
  The Core Outcome Measurement Index consists of seven items that assess pain, neck-related function, symptom-specific well-being, general quality of life, and disability. Except for the questions about the patient's disability in the previous 4 weeks, all questions are about how the patient felt in the previous week. Increasing score indicates worse condition.
General quality of life assessed by Nottingham Health Profile | 1 day
  The Nottingham Health Profile is a general quality of life questionnaire that measures a person's perceived health problems and the extent to which these problems affect normal daily activities. The questionnaire consists of 38 items. Questions are answered as 'yes' or 'no'. The questionnaire assesses six parameters related to health status. These parameters are; pain (8 items), physical activity (8 items), energy (3 items), sleep (5 items), social isolation (5 items), and emotional reactions (9 items). Each subparameter is scored between 0-100. 0 indicates best health, and 100 indicates worst health. The total NHP score is derived from the sum of the subscores.
Japanese Orthopedic Association Back Pain Evaluation Questionnaire | 1 day
  The Japanese Orthopedic Association Back Pain Evaluation Questionnaire is a disease-specific self-assessment questionnaire for back pain. It consists of five subscales (social function, mental health, low back function, walking ability and low back pain) and 25 items. Each subscale score ranges from 0 to 100. Higher scores indicate better conditions.
The Bournemouth Questionnaire | 1 day
  The Bournemouth Questionnaire is a multidimensional scale that evaluates pain, daily-social life, depression-anxiety, pain control and fear avoidance behaviors with seven questions. Increasing score indicates worse condition.
The Spine Functional Index | 1 day
  The Spine Functional Index is a 25-item questionnaire completed according to the patient's functional status in the "last few days". Scores from 25 items are added together, then this score is multiplied by four and subtracted from 100 to obtain a percentage score. Increasing score indicates worse condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Merkez, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No